CLINICAL TRIAL: NCT03976856
Title: A Phase Ib Clinical Study With Extension Phase to Evaluate Safety and Efficacy of Genolimzumab (GB226) in Combination With Fruquintinib in the Treatment of Relapsed or Metastatic NSCLC Patients
Brief Title: Safety and Efficacy of Genolimzumab (GB226) in Combination With Fruquintinib
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Collaborators: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gxplore-015
Record Dates: First submitted 2019-05-24; First posted 2019-06-06 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GB226+Fruquintinib (Experimental): Geptanolimab combined with Fruquintinib
  Interventions: Drug: GB226; Drug: Fruquintinib

INTERVENTIONS:
Drug: GB226 — Geptanolimab, 210mg，q2w，ivgtt.
  Other Names: Geptanolimab
Drug: Fruquintinib — Fruquintinib, 3mg or 4mg or 5mg, qd.po. 3 weeks-on,1 week-off
  Other Names: HMPL-013

SUMMARY:
This study is a multi-center, open-label, dose-finding phase Ib clinical study with extension phase, which is aimed at evaluating the efficacy and safety of GB226 combined with fruquintinib in treatment of relapsed or metastatic NSCLC patients with EGFR-sensitive mutations who have failed to respond to EGFR-TKI treatment,evaluating the pharmacokinetic characteristics of GB226 and fruquintinib, and the immunogenicity of GB226, and preliminarily evaluating the antitumor activity of GB226 and fruquintinib.

DETAILED DESCRIPTION:
In this study, it is planned to enroll at least 42 NSCLC patients who meet relevant criteria. This study includes dose escalation phase and extension phase of the combined therapy: three combined dose groups are planned in the dose escalation phase; the dose extension phase is divided into two cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, male or female;
2. Understanding the procedures and contents of the study, and voluntarily signing the written informed consent form;
3. Histologically or cytology confirmed relapsed or metastatic NSCLC;
4. EGFR gene sensitive mutation is confirmed positive, any of following is met: exon 19 deletion (19DEL), exon 21 point mutation (L858R / L861Q), 18 exon point mutation (G719X), 20 exon point mutation (S768I). Moreover, the following conditions are met:

   1. No T790M mutation after failure of EGFR-TKI treatment;
   2. T790M mutation after EGFR-TKI treatment failure, and failed to respond to third-generation EGFR-TKI treatment; primary T790M mutation, progressed after third-generation EGFR-TKI treatment or no other available effective therapies;
   3. The above patients failed to respond to chemotherapy or are unwilling to or intolerable to chemotherapy;
5. According to the RECIST 1.1 criteria, at least one target lesion (the lesion with a longest diameter ≥10 mm, or a lymph node with a short diameter ≥15 mm) are measured by CT or MRI;
6. Expected survival ≥ 3 months;
7. ECOG score: 0-1;
8. Completion of systemic chemotherapy, radical/extensive therapy, or previous anti-tumor biological therapies (tumor vaccine, cytokine or growth factor for the purpose of tumor control) for at least 4 weeks, completion of local palliative radiotherapy for at least 1 week;
9. The EGFR-TKI treatment has ended over 2 weeks before the use of study drugs;
10. Patients who have not previously received treatment with TKI or monoclonal antibodies against Vascular Endothelial Growth Factor (VEGF) and/or VEGFR;
11. At least 8 weeks after completion of major surgery requiring general anesthesia before the use of study drugs; at least 4 weeks after completion of surgery requiring local anesthesia/epidural anesthesia and recovery from the surgery;
12. Discontinuation of systemic corticosteroids for at least 2 weeks before the use of study drugs (prednisone > 10 mg/day or equivalent dose);
13. The values of the laboratory tests performed for screening must meet the following criteria:

    Blood routine test results(no blood transfusion, G-CSF or other drugs for correction within 14 days before screening):
    1. Hemoglobin HGB ≥90g/L;
    2. Absolute neutrophil count (ANC) ≥1.5x10^9/L;
    3. Platelet count PLT ≥100x10^9/L;

    Clinical biochemistry:
    1. Total bilirubin (TBIL) ≤1.5 times the upper limit of normal [ULN] [≤1.5 times for Gilbert syndrome);
    2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times the ULN (AST and/or ALT ≤5×ULN for patients with liver metastases);
    3. Serum creatinine ≤ 1.5 × ULN or endogenous creatinine clearance rate≥ 50 mL/min (Cockcroft-Gault formula)
    4. Urine protein ˂ 2+ or ˂1.0 g/L. For patients with baseline urinary protein ≥ 2+ or ≥ 1.0 g/L, a 24-hour urine protein quantitative test should be performed, and the result should be ≤ 1.0 g/L;

    Coagulation Function:

    a)Activated partial thromboplastin time (APTT) or prothrombin time (PT) ≤1.5 times ULN
14. Thyroid function variables: thyroid stimulating hormone (TSH), free thyroxine (FT3/FT4) within the normal range;
15. Recovery of adverse reactions caused by previous treatment to grade 1 and below before enrollment (except hair loss and ≤grade 2 neurotoxicity caused by chemotherapeutic agents);
16. Women who are confirmed not pregnant within within 7 days before administration; male or female subjects who are able to father or bear a child agree to take medically recognized effective contraceptive measures throughout the study period and within six months of completion of the study;
17. Consent to provide tissue samples and receive biopsy if necessary.

Exclusion Criteria:

1. Patients with lung squamous cell carcinoma (including adenosquamous carcinoma);
2. ALK fusion gene rearrangement confirmed by genetic testing;
3. Patients with history of other malignant tumors (except cured cervical carcinoma in situ, basal cell carcinoma of skin or squamous cell carcinoma) may not participate in the study unless the diseases have been cured for at least 5 years prior to enrollment, and it is estimated that no other treatment will be required throughout the study;
4. Detection of the tumor lesion ≤ 5 mm from the large vessel, or a central tumor that invaded the local large vessel; or a significant pulmonary cavity or necrotizing tumor by imaging (CT or MRI);
5. Active central nervous system (CNS) metastasis, including symptomatic brain metastasis, meningeal metastasis or spinal cord compression; patients with asymptomatic brain metastases can be enrolled (no progression and/or neurological symptoms or signs after surgical resection within at least 4 weeks after radiotherapy, no history of treatment with glucocorticoids, anticonvulsants or mannitol);
6. Symptomatic, uncontrollable serous effusions such as ascites, pleural effusion, or pericardial effusion;
7. History of arterial thrombosis or deep vein thrombosis within 6 months prior to enrollment, evidence or history of bleeding tendency within 2 months prior to enrollment, regardless of severity;
8. Patients with thrombolytic therapy or therapeutic anticoagulant drugs (except prophylactic anticoagulant drugs) within 10 days before the first study drug;
9. History of active, known autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, except type I diabetes, hypothyroidism that can be controlled by hormone replacement therapy only, skin diseases not requiring systemic treatment (such as vitiligo and psoriasis) and controlled celiac disease.
10. Previous treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibodies (or any other antibodies that act on T-cell costimulatory or checkpoint pathways);
11. Uncontrolled hypertension (systolic blood pressure﹥140mmHg and/or diastolic blood pressure﹥90mmHg), pulmonary hypertension or unstable angina; myocardial infarction, bypass surgery or stent surgery within 6 months before administration of drug; history of chronic heart failure that meets the criteria for grade 3-4 defined by New York Heart Association (NYHA); severe arrhythmia requiring treatment, including QTc interval ≥450ms for male subjects and ≥ 470ms for female subjects (calculated by Fridericia formula); left ventricular ejection fraction (LVEF) <50%; cerebral vascular accident (CVA) or transient ischemic attack (TIA) within 6 months before administration of drug;
12. Skin wounds, surgical site, wound site, severe mucosal ulcers or fractures that are not completely healed;
13. Dysphagia or gastrointestinal disorders that may significantly affect absorption of oral drugs or any conditions that may cause gastrointestinal bleeding or perforation at the discretion of the investigator (such as duodenal ulcer, gastrointestinal obstruction, diverticulitis, intraperitoneal abscess, metastasis of peritoneal carcinoma, acute Crohn's disease, ulcerative colitis, large area stomach and small bowel resection). Patients with chronic Crohn's disease and ulcerative colitis (except total colon and rectal resection) should be excluded even during inactivity period. Patients with hereditary nonpolyposis colorectal cancer or familial adenomatous polyposis syndrome; patients with history of intestinal perforation and intestinal fistula who are not recovered after surgery;
14. Previouly or currently suffered from active tuberculosis infection, or other infections requiring systemic treatment;
15. Positive human immunodeficiency virus antibody (HIV-Ab), treponema pallidum antibody (TP-Ab) or hepatitis C antibody (HCV-Ab); positive hepatitis B virus surface antigen (HBsAg), and hepatitis B virus DNA copy number > upper limit of normal of the testing institution;
16. Complications requiring treatment with immunosuppressive drugs or requiring systemic use of doses with immunosuppressive effects (prednisone >10 mg/day or equivalent dose of similar drugs); in the absence of active autoimmune disease, it is allowed to inhale or topically use steroids and prednisone >10mg/day or similar drugs at an equivalent dose.
17. History of interstitial lung disease;
18. Received treatment with other study drugs within 30 days before administration of the study drug or before 5 half-lives of other study drugs (whichever is longer); or use of investigational device within 30 days;
19. Live vaccines or attenuated vaccines are expected to be administered within 4 weeks before administration, during treatment period or within 5 months after the last dose;
20. History of drug addiction or drug abuse upon inquiry;
21. Breastfeeding women;
22. Known allergy to recombinant humanized PD-1 monoclonal antibody or any of its excipients; known allergy to analogues of fruquintinib; known history of allergic diseases or severe allergic constitution;
23. Other circumstances based on which the investigator believes that the subject is not suitable for participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Event | all adverse events will be recorded from the time the consent form is signed through 90 days following cessation of treatment.
  Assessment of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Incidence of Serious Adverse Event | all adverse events will be recorded from the time the consent form is signed through 90 days following cessation of treatment.
  Assessment of serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Dose Limited Toxicity | Day 1 to Day 28 after first dose
  Incidence of Dose Limited Toxicity
Maximum Tolerated Dose | Day 1 to Day 28 after first dose
  Defined as the highest dose tested in which only 0 or 1 out of 6 evaluable patients experience a dose limiting toxicity, as graded by the National Cancer Institute (NCI) Common terminology Criteria for Adverse Events (CTCAE) version 4.03

SECONDARY OUTCOMES:
Cmax | up to 90 days after the last administration
  Cmax
Tmax | up to 90 days after the last administration
  Tmax
AUC0-t | up to 90 days after the last administration
  AUC0-t
AUC0-∞ | up to 90 days after the last administration
  AUC0-∞
MRT | up to 90 days after the last administration
  MRT
Vd | up to 90 days after the last administration
  Vd
CL | up to 90 days after the last administration
  CL
AUC 0-τ | up to 90 days after the last administration
  AUC 0-τ
C avg | up to 90 days after the last administration
  C avg
C min | up to 90 days after the last administration
  C min
CL ss | up to 90 days after the last administration
  CL ss
Objective Response Rate, ORR | up to 90 days after the last administration
  To evaluate the efficacy of GB226 as defined by objective response rate in patients with lung cancer.
Disease control rate,DCR | up to 90 days after the last administration
  To evaluate the efficacy of GB226 as defined by disease control rate in patients with lung cancer.
Duration of response, DOR | up to 90 days after the last administration
  To evaluate the duration of response (DOR) of GB226 in patients with lung cancer
Progression-free survival, PFS | up to 90 days after the last administration
  To evaluate the efficacy of GB226 as defined by progression-free survival in patients with lung cancer
Overall survival, OS | up to 90 days after the last administration
  To evaluate the efficacy of GB226 as defined by overall survival in patients with lung cancer.
Concentration of AntiDrug Antibody, ADA | up to 90 days after the last administration
  To evaluate the immunogenicity of GB226 in Chinese patients with lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Doctor, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai chest hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No